CLINICAL TRIAL: NCT06948890
Title: Effect of Music on Cue Reactivity for Patients With Opioid Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Scott G. Weiner, MD, MPH, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025P000151
Record Dates: First submitted 2025-04-20; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Opioid Use Disorder
Keywords: opioid; opioid use disorder; methadone; buprenorphine; music; cue reactivity
MeSH Terms: conditions — Opioid-Related Disorders | interventions — SIR1 protein, S cerevisiae

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music (Experimental): In this arm, subjects will rate their cravings for opioids on a 0-100 point visual analog scale. They will then listen to 2 songs of their choosing. They will then be shown a series of images "cues" related to drug use, and will again be asked their cravings for opioids.
  Interventions: Other: Music intervention
- silence (Placebo Comparator): In this arm, subjects will rate their cravings for opioids on a 0-100 point visual analog scale. They will then listen to 10 minutes of silence. They will then be shown a series of images "cues" related to drug use, and will again be asked their cravings for opioids.
  Interventions: Other: Silence

INTERVENTIONS:
Other: Music intervention — Subjects will listen to two songs of their choosing. They will be prompted: "Please choose two songs that you really enjoy and that make you feel relaxed or take away stress".
  Arms: music
Other: Silence — Subjects will listen to 10 minutes of silence through high quality noise canceling headphones
  Arms: silence

SUMMARY:
This research is being performed to understand the role of music in people's opioid cravings, opioid use, and recovery. Music affects individuals in so many ways, and can trigger strong good and bad emotions. People listen when they are sad and want to feel happy, when they are with friends, when they exercise, and when they just want to pass the time. However, it is not known what role music plays in adding to or taking away cravings, and the role it has in drug use and addiction. In this study, the researchers want to learn if music can reduce cues that lead to cravings for opioids. The researchers also want to learn about subjects' relationship to music and how it contributes to drug use, recovery, and their life overall.

DETAILED DESCRIPTION:
Opioid use disorder (OUD) presents a significant public health challenge, characterized by a complex interplay of biological, psychological, and environmental factors. One critical aspect of this disorder is cue reactivity, the phenomenon whereby exposure to drug-related cues trigger cravings and reinforce behaviors to use drugs. This study aims to explore the role of music as a potential modulator of cue reactivity in patients with OUD.

Music, with its profound emotional and psychological effects, may offer a unique avenue for intervention. Previous research has demonstrated that music can influence mood, reduce anxiety, and enhance emotional regulation. Listening to music may also attenuate nociceptive processing and change thresholds of pain tolerance. By examining how specific musical stimuli interact with drug-related cues, the researchers hope to identify whether music can serve as an adjunctive strategy or an emotional anchor that diminishes cravings associated with opioid cues. This research seeks to contribute to the development of innovative therapeutic strategies aimed at reducing relapse rates and promoting recovery among individuals struggling with OUD.

Through a carefully designed mixed methods experimental framework, the researchers will assess the effects of different musical genres on cue-induced cravings. It is anticipated that the findings will provide valuable insights into the potential of music as a complementary tool in the treatment of opioid use disorder, paving the way for more holistic and effective recovery approaches.

Specific Aim 1: To determine the effect of music on cue-induced craving for individuals with opioid use disorder compared to a control condition (silence).

Hypothesis 1: Compared to the control condition, listening to music will attenuate cue-induced craving as assessed on a 100-point VAS craving scale.

Specific Aim 2: Identify the role of music in people's use of opioids through individual interviews with study participants.

Hypothesis 2: There will be key themes that emerge related to people's use of opioids as well as in their treatment and recovery.

This is a donor-funded, open label, pilot, proof-of-concept study with two parts. The study will aim to randomize N=28 individuals (14 in control arm and 14 in intervention arm) who have a history of opioid use disorder. Individuals will be recruited from a variety of means including online study recruitment and through fliers stationed at MGB-affiliated addiction clinics (including the Brigham and Women's Hospital and Massachusetts General Hospital Bridge Clinics, the Faulkner Addiction Recovery Program, and the MGH West End clinic).

Participants who agree to participate in the study will come to the Center for Clinical Investigation (CCI) once. The entirety of the study for each participant entails one CCI visit.

In the first phase, participants will answer a demographic questionnaire and a variety of psychological assessments. They will answer a question pertaining to their degree of opioid craving at that moment, on a 100-point visual analog scale (VAS). They will then be randomized to listen to music (2 songs chosen by them, maximum 10 minutes) or 10 minutes of noise cancelation. Participants will then be shown a series of images related to opioid use. They will complete the craving scale again. They will be shown a series of neutral images that do not pertain to drug use, and the craving scale will be administered again. Finally, they will complete the Absorption in Music Scale.

The second phase, for all participants regardless of randomization in the first phase, will be a qualitative interview asking subjects about their relationship with music, and how music pertained to their past drug use and/or recovery. Researchers will also ask participants about their experience participating in the trial and potential strategies to expand music use and recommendations in clinical settings for OUD.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Current diagnosis of opioid use disorder
* Actively receiving buprenorphine or methadone treatment with a stable dose of at least 30 days

Exclusion Criteria:

* Any significant impairment in mental status that would interfere with the ability to provided informed consent including suicidality, homicidality, or psychosis.
* Hearing impaired
* Vision impaired
* Patient reports that they are pregnant
* Requiring the use of any prescription opioid analgesics during the trial
* Currently prescribed naltrexone
* Chronic pain, defined as pain on the numeric rating scale (0-10) of >3 every day for over 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Opioid Cravings | on Day 1
  Subjects will rank their craving for opioids on a 100-point Visual Analog Scale before and after being shown drug-related cues (images). The primary outcome will determine if there is a difference in craving levels in the music vs. silence groups.

CONTACTS AND LOCATIONS:
Overall Officials: Scott G Weiner, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suzuki J, Martin B, Prostko S, Chai PR, Weiss RD. Cannabidiol Effect on Cue-Induced Craving for Individuals with Opioid Use Disorder Treated with Buprenorphine: A Small Proof-of-Concept Open-Label Study. Integr Med Rep. 2022 Aug 1;1(1):157-163. doi: 10.1089/imr.2022.0070. Epub 2022 Aug 26. PMID 36105269
- [Background] Chai PR, Carreiro S, Ranney ML, Karanam K, Ahtisaari M, Edwards R, Schreiber KL, Ben-Ghaly L, Erickson TB, Boyer EW. Music as an Adjunct to Opioid-Based Analgesia. J Med Toxicol. 2017 Sep;13(3):249-254. doi: 10.1007/s13181-017-0621-9. Epub 2017 Jun 23. PMID 28646359
- [Background] Chai PR, Schreiber KL, Taylor SW, Jambaulikar GD, Kikut A, Hasdianda MA, Boyer EW. The Feasibility and Acceptability of a Smartphone-Based Music Intervention for Acute Pain. Proc Annu Hawaii Int Conf Syst Sci. 2019 Jan 8;2019:3917-3925. PMID 30700971
- [Background] Chai PR, Schwartz E, Hasdianda MA, Azizoddin DR, Kikut A, Jambaulikar GD, Edwards RR, Boyer EW, Schreiber KL. A Brief Music App to Address Pain in the Emergency Department: Prospective Study. J Med Internet Res. 2020 May 20;22(5):e18537. doi: 10.2196/18537. PMID 32432550
- [Background] Colebaugh CA, Wilson JM, Flowers KM, Overstreet D, Wang D, Edwards RR, Chai PR, Schreiber KL. The Impact of Varied Music Applications on Pain Perception and Situational Pain Catastrophizing. J Pain. 2023 Jul;24(7):1181-1192. doi: 10.1016/j.jpain.2023.01.006. Epub 2023 Jan 14. PMID 36646399
- See also: Related Info — https://rally.massgeneralbrigham.org/study/musicoud